CLINICAL TRIAL: NCT06924372
Title: Application of Salivary Biomarkers in Risk Assessment for Oral Diseases in Children With Type 1 Diabetes
Status: Active, not recruiting | Type: Observational
Sponsor: University of Novi Sad (Other)
Responsible Party: Principal Investigator, Bojan Petrovic, Full professor at University of Novi Sad, Medical faculty, University of Novi Sad
Other Study IDs: Number:01-17/13-2023
Record Dates: First submitted 2025-04-02; First posted 2025-04-11 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2025-04

CONDITIONS: Biomarkers; Saliva; Type 1 Diabetes (T1D); Dental Care for Children
Keywords: salivary biomarkers; type 1 diabetes T1D; children; oral disease
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Mouth Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Experimental group: Age of subjects from 6 to 18 years, both sexes, with mixed or permanent dentition present. An experimental group of at least 56 subjects will be children diagnosed with DM type 1 (at least one year), who are treated at the Novi Sad Health Center, Children's Health Care Service, and will be referred to the Department of Pediatric and Preventive Dentistry, Clinic for Dentistry of Vojvodina. The experimental group will be divided into two subgroups: at least 28 subjects with well-regulated type 1 DM and at least 28 subjects with poorly regulated type 1 DM.
  Interventions: Other: Taking saliva samples of unstimulated saliva will be collected in sterile containers, salivets.; Other: Dental status; Other: Periodontal status
- Control group: The control group includes at least 56 subjects, healthy children, who match the tested group in gender and age, patients of the Clinic of Dentistry of Vojvodina, with the absence of acute diseases. Age of subjects from 6 to 18 years, both sexes, with mixed or permanent dentition present.
  Interventions: Other: Taking saliva samples of unstimulated saliva will be collected in sterile containers, salivets.; Other: Dental status; Other: Periodontal status

INTERVENTIONS:
Other: Taking saliva samples of unstimulated saliva will be collected in sterile containers, salivets. — Subjects will sit in a filiological position in a dental chair. Samples of unstimulated saliva will be collected in sterile containers, salivets. A prerequisite for taking saliva samples will be that subjects do not take water and food until two hours before the examination, according to the manufacturer's instructions. SARSTED Salivette will be used. In a sterile manner, the swab will be removed from the salivette with sterile tweezers and applied to the patient's mouth on the buccal mucosa. The tampon will be held for a minimum of 2 minutes in the patient's mouth (with buccal mucosa). After the elapsed time, the tampon will be removed from the mouth, using sterile tweezers and sterile gloves and will be inserted into the saliva and closed. After sampling, the salivates will be transported to the Department of Microbiological Diagnostics of the Institute for Pulmonary Diseases of Vojvodina. Transport should be done in the shortest possible time.
Other: Dental status — Dental status in both groups of subjects will be assessed by clinical visual examination by determining the prevalence of caries of deciduous and permanent teeth using the KEP and KEPS indexes. The clinical examination will be carried out in a dental chair using artificial light-reflectors, using a dental mirror and a dental probe on all surfaces of the tooth, which are dried with air from the puster. On the basis of a dental examination, the prevalence of caries of deciduous and permanent teeth will be determined.
Other: Periodontal status — The assessment of the presence of dental plaque will be determined visually using the Silness and Loe plaque index, while the condition of the gingiva will be determined using the gingival index Loe and Silness . Before the examination, the subject will be advised to rinse his mouth with water to remove food residues and dental plaque. Performed in the dental chair using artificial light-reflectors, by gently pulling the dental probe over the vestibular, oral, mesial and distal surfaces of all crowns of the present teeth. Four values will be entered for each tooth. The result will be obtained by adding up all the values.

SUMMARY:
This research contributes to a deeper understanding of the etiopathogenesis of periodontal and other oral diseases in children with T1D. By analyzing the composition of the salivary microbiome and detecting pathogenic and opportunistic microorganisms, the study aims to develop targeted preventive strategies. The findings could lead to personalized preventive programs, improving early diagnosis and oral health management in this vulnerable population.This study hypothesizes that children with Type 1 Diabetes (T1D) will exhibit significantly different oral health parameters compared to healthy peers. Specifically:

1. Higher KEP and KEPS index values (Klein-Palmer system) indicating increased caries incidence.
2. Higher Silness and Loe plaque index and Loe and Silness gingival index, suggesting greater plaque accumulation and gingival inflammation.
3. Lower salivary buffering capacity and pH, potentially contributing to an increased risk of oral diseases.
4. A distinct microbial profile, with a greater presence of pathogenic and opportunistic bacteria.
5. A significantly higher Candida albicans count in the saliva. These findings could provide insights into the oral health challenges faced by children with T1D and guide preventive strategies.

This study explores how saliva can help assess the risk of dental and gum problems in children with Type 1 Diabetes (T1D). Researchers will analyze saliva samples to identify specific markers that may indicate a higher chance of cavities, gum disease, and oral infections. The goal is to develop early detection and prevention methods to improve oral health care for children with T1D.

The study will include 112 children aged 6 to 18. Half of them have Type 1 Diabetes, while the other half are healthy children of the same age and gender for comparison. All participants will be selected from the Clinic for Dentistry of Vojvodina, ensuring they are not currently sick and have not taken antibiotics in the past month. Children with other serious health conditions, fixed braces, or difficulty cooperating will not be included.

Researchers will examine different factors that could affect oral health in children with T1D, including saliva acidity (pH), its ability to neutralize acids, the presence of bacteria and fungi, and the condition of teeth and gums. They expect that children with T1D will have:

1. More cavities compared to healthy children.
2. More plaque buildup on teeth and greater gum inflammation.
3. Lower saliva protection against acids, increasing the risk of dental problems.
4. A different mix of bacteria in the mouth, with more potentially harmful microbes.
5. Higher levels of the fungus Candida albicans in saliva. The findings from this study may help better understand oral health challenges in children with T1D and lead to improved prevention and treatment strategies.

DETAILED DESCRIPTION:
Diabetes mellitus (DM) is a metabolic disorder characterized by impaired metabolism of carbohydrates, fats, and proteins. As a chronic disease, it leads to numerous systemic complications (1). Type 1 diabetes mellitus (T1DM) most commonly affects children and adolescents, although it may also occur in adults, potentially due to modern lifestyle factors (2). The incidence and prevalence of T1DM are increasing globally, posing a significant public health and economic burden. In response, preventive programs are being developed to reduce the impact of diabetes in the general population (3). Typical symptoms of T1DM in children include frequent nocturnal urination, increased thirst, unexplained weight loss, constant hunger, hyperglycemia, blurred vision, and extreme fatigue. Additional signs may include abdominal pain, shortness of breath, or vomiting (4). In younger children, T1DM is associated with a heightened risk of diabetic ketoacidosis-the most severe and life-threatening complication of T1DM-as well as a greater risk of microvascular and macrovascular complications, often resulting in hospitalization (5).

Children and adolescents with T1DM experience absolute insulin deficiency and require lifelong exogenous insulin therapy. Treatment focuses on achieving glycemic control and preventing complications through a combination of dietary management, physical activity, and insulin therapy-delivered either via intensified insulin regimens or insulin pumps. This approach also requires frequent monitoring, regular clinical check-ups, and high levels of education and engagement from both patients and their parents (3).

The oral cavity is frequently affected by T1DM (3). Individuals with diabetes commonly experience oral health issues such as impaired taste, periodontal disease, salivary gland dysfunction, sensory disturbances, and an increased susceptibility to dental caries and oral infections (6). The properties of saliva play a crucial role in maintaining oral health and preventing caries. Saliva protects the oral tissues, provides a defense mechanism against bacteria, fungi, and viruses (7), and regulates demineralization and remineralization processes in the cariogenic environment (8). Its buffering capacity stabilizes oral pH, thereby helping to prevent enamel demineralization (8).

Insulin deficiency in T1DM leads to both qualitative and quantitative alterations in saliva, including hyposalivation and elevated salivary glucose concentrations. These changes are associated with a higher risk of caries and periodontal disease (9). Several key factors influence the development of caries, including frequent consumption of fermentable carbohydrates, poor oral hygiene, reduced fluoride intake, and the biological characteristics of saliva (10). Studies have reported increased counts of Streptococcus mutans and Lactobacillus spp. in individuals with T1DM, particularly in those with poor metabolic control, potentially due to elevated glucose levels in saliva and gingival crevicular fluid (9,11). The relationship between T1DM and periodontal health is well established. Children with T1DM, especially those with poor glycemic control, are at increased risk of developing chronic gingivitis, which tends to worsen with age (10-12). Glycosylated hemoglobin A1c (HbA1c) is a key marker used to evaluate average blood glucose levels over the preceding two to three months. The American Diabetes Association (ADA) recommends measuring HbA1c levels three to four times per year in patients with T1DM to assess metabolic control (13). According to ADA guidelines, good metabolic control in school-aged children (6-12 years) is defined by an HbA1c level <8%, while for adolescents and young adults (13-19 years), the target is <7.5%.

Studies examining the oral microbiota have shown significant differences between children with T1DM and healthy children. Notably, higher counts of periodontal pathogens, S. mutans, and Lactobacillus have been documented in children with T1DM (10-12). Reports on Candida albicans are mixed: while some studies show no significant difference, others suggest higher prevalence in children with T1DM compared to healthy controls (10). These discrepancies highlight the need for further research to clarify the impact of T1DM on the oral microbiota. Previous research has linked poor metabolic control in T1DM with increased risk for oral diseases. Risk assessment has traditionally included measures of caries prevalence, salivary flow rate, buffering capacity, and bacterial counts in stimulated saliva (11). Beyond its protective role, saliva also serves as a valuable diagnostic tool for both oral and systemic diseases. Saliva collection is simple, painless, and non-invasive, making it ideal for clinical and research use (14). Identifying reliable salivary biomarkers could contribute to the prevention, diagnosis, and prognosis of oral diseases in children with T1DM (15). Mass spectrometry (MS) has emerged as a powerful technique for comprehensive salivary proteomic analysis. It enables quantitative mapping of both host and microbial proteins in saliva (16). This highly sensitive method can identify both known and novel compounds and is increasingly applied in dental and biomedical research (17,18).

The findings from this study aim to deepen our understanding of the oral microbiota in children with T1DM and its diagnostic potential in oral disease development. By identifying specific salivary biomarkers, particularly through the use of MS, it may be possible to predict and prevent oral diseases in this vulnerable population. These insights could support the development of personalized preventive and prophylactic programs, improving both oral health and overall quality of life in children with T1DM. Ultimately, this research may help pediatric dentists tailor their clinical and preventive care to reduce the risk of oral complications in children with type 1 diabetes, while also advancing the broader understanding of the relationship between T1DM and oral health.

ELIGIBILITY:
Inclusion Criteria:

* Age of subjects from 6 to 18 years, both sexes, with mixed or permanent dentition present.
* An experimental group of at least 56 subjects will be children diagnosed with DM type 1 (at least one year)
* The control group includes at least 56 subjects, healthy children, who match the tested group in gender and age, with the absence of acute diseases.

Exclusion Criteria:

* Uncooperative patient
* Associated diseases
* Unsigned informative consent from the data subject/parent/guardian
* Antibiotic use in the last few months
* Subjects with orthodontic appliances

Ages: 6 Years to 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: An experimental group will be children diagnosed with DM type 1 (at least one year), who are treated at the Novi Sad Health Center, Children's Health Care Service, and will be referred to the Department of Pediatric and Preventive Dentistry, Clinic for Dentistry of Vojvodina.
  The control group includes healthy children, who match the tested group in gender and age, patients of the Clinic of Dentistry of Vojvodina
Sampling Method: Non-Probability Sample
Enrollment: 112 (Estimated)
Dates: Start 2025-01-31 (Actual); Primary Completion 2025-07-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Prevalence of dental caries and periodontal disease | From 31 January 2025 to January 2026
  The primary outcome of the study is the prevalence of dental caries and periodontal diseases in children with type 1 diabetes, compared to non-diabetic children. Caries prevalence will be defined using KEP and KEPS indexes according to the Klein-Palmer system and assessment of the amount of dental plaque using the Silness and Loe plaque index and assessment of gingival condition using the gingival index Loe and Silness .
Microbiological analysis | From 31 January 2025 to January 2026
  The primary outcome of this clinical research is to evaluate the feasibility and effectiveness of collecting unstimulated saliva samples for microbiological procedures and analysis. Specifically, the study aims to determine whether unstimulated saliva can serve as a reliable diagnostic medium for the identification and characterization of isolated microorganisms present in the oral cavity. The identification of these microorganisms will be carried out using standard microbiological techniques to assess the microbial composition and potential pathogenic species. Outcomes will be measured based on data provided after experimental part.

SECONDARY OUTCOMES:
Saliva chek buffer | From 31 January 2025 to January 2026.
  Evaluation of the characteristics of stimulated saliva - buffering capacity of saliva in children with DM type 1 and healthy subjects.
  Invitro test for cheking buffering capacity of saliva using saliva from collection cup. Final results will be calculated by adding the points from 0-12 according to the final colour of each pad.
Saliva ph measurement | From 31 January 2025 to January 2026
  In vitro test for ph measurement of saliva. According to the manufacturer's instructions using ph test strip and pooled saliva expectorated in the collection cup. Measuring the pH value of saliva using a factory-made color scale and determining the pH of saliva on a scale from 5.0 to 7.8.

OTHER OUTCOMES:
Questionnaire | From 31 January 2025 to January 2026
  Oral health related quality of life, as reported through validated questionnaires or surveys in studies, to assess how dental caries and diabetes management affect overall well-being.
  Outcomes will be measured based on data provided after experimental part. Measures of effect.

CONTACTS AND LOCATIONS:
Locations (1):
- Medical Faculty, University of Novi Sad, Novi Sad, Serbia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Ziegler R, Neu A. Diabetes in Childhood and Adolescence. Dtsch Arztebl Int. 2018 Mar 2;115(9):146-156. doi: 10.3238/arztebl.2018.0146. PMID 29563012
- [Background] Petrovic B, Stilinovic N, Tomas A, Kojic S, Stojanovic GM. Determination of salivary concentrations of leptin and adiponectin, ability to reduce ferric ions and total antioxidant capacity of saliva in patients with severe early childhood caries. Front Pediatr. 2022 Aug 31;10:969372. doi: 10.3389/fped.2022.969372. eCollection 2022. PMID 36120658
- [Background] 16. Nirmala SVSG, Saikrishna D. Dental Care and Treatment of Children with Diabetes Mellitus- An Overview. J Pediatr Neonatal Care.2016; 4(2): 00134.
- [Background] Chi LM, Hsiao YC, Chien KY, Chen SF, Chuang YN, Lin SY, Wang WS, Chang IY, Yang C, Chu LJ, Chiang WF, Chien CY, Chang YS, Chang KP, Yu JS. Assessment of candidate biomarkers in paired saliva and plasma samples from oral cancer patients by targeted mass spectrometry. J Proteomics. 2020 Jan 16;211:103571. doi: 10.1016/j.jprot.2019.103571. Epub 2019 Nov 2. PMID 31689561
- [Background] Kallianta M, Pappa E, Vastardis H, Rahiotis C. Applications of Mass Spectrometry in Dentistry. Biomedicines. 2023 Jan 19;11(2):286. doi: 10.3390/biomedicines11020286. PMID 36830822
- [Background] Ahmad P, Hussain A, Siqueira WL. Mass spectrometry-based proteomic approaches for salivary protein biomarkers discovery and dental caries diagnosis: A critical review. Mass Spectrom Rev. 2024 Jul-Aug;43(4):826-856. doi: 10.1002/mas.21822. Epub 2022 Nov 29. PMID 36444686
- [Background] 12. Classification and Diagnosis of Diabetes: Standards of Care in Diabetes-2023.Diabetes Care 2023; 46 (Suppl. 1): S19-S40.
- [Background] Rapone B, Corsalini M, Converti I, Loverro MT, Gnoni A, Trerotoli P, Ferrara E. Does Periodontal Inflammation Affect Type 1 Diabetes in Childhood and Adolescence? A Meta-Analysis. Front Endocrinol (Lausanne). 2020 May 5;11:278. doi: 10.3389/fendo.2020.00278. eCollection 2020. PMID 32431669
- [Background] Mohamed HG, Idris SB, Mustafa M, Ahmed MF, Astrom AN, Mustafa K, Ibrahim SO. Influence of Type 2 Diabetes on Prevalence of Key Periodontal Pathogens, Salivary Matrix Metalloproteinases, and Bone Remodeling Markers in Sudanese Adults with and without Chronic Periodontitis. Int J Dent. 2016;2016:6296854. doi: 10.1155/2016/6296854. Epub 2016 Feb 17. PMID 26989414
- [Background] Novotna M, Podzimek S, Broukal Z, Lencova E, Duskova J. Periodontal Diseases and Dental Caries in Children with Type 1 Diabetes Mellitus. Mediators Inflamm. 2015;2015:379626. doi: 10.1155/2015/379626. Epub 2015 Aug 4. PMID 26347009
- [Background] Animireddy D, Reddy Bekkem VT, Vallala P, Kotha SB, Ankireddy S, Mohammad N. Evaluation of pH, buffering capacity, viscosity and flow rate levels of saliva in caries-free, minimal caries and nursing caries children: An in vivo study. Contemp Clin Dent. 2014 Jul;5(3):324-8. doi: 10.4103/0976-237X.137931. PMID 25191067
- [Background] Dabelea D. The accelerating epidemic of childhood diabetes. Lancet. 2009 Jun 13;373(9680):1999-2000. doi: 10.1016/S0140-6736(09)60874-6. Epub 2009 May 27. No abstract available. PMID 19481250
- [Background] Ferizi L, Dragidella F, Spahiu L, Begzati A, Kotori V. The Influence of Type 1 Diabetes Mellitus on Dental Caries and Salivary Composition. Int J Dent. 2018 Oct 2;2018:5780916. doi: 10.1155/2018/5780916. eCollection 2018. PMID 30369949
- [Background] Nazir MA, AlGhamdi L, AlKadi M, AlBeajan N, AlRashoudi L, AlHussan M. The burden of Diabetes, Its Oral Complications and Their Prevention and Management. Open Access Maced J Med Sci. 2018 Aug 15;6(8):1545-1553. doi: 10.3889/oamjms.2018.294. eCollection 2018 Aug 20. PMID 30159091
- [Background] Ferizi L, Bimbashi V, Kelmendi J. Association between metabolic control and oral health in children with type 1 diabetes mellitus. BMC Oral Health. 2022 Nov 16;22(1):502. doi: 10.1186/s12903-022-02555-x. PMID 36384715
- [Background] Assiri SA, El Meligy OAES, Alzain IO, Bamashmous NO. Assessment of dental caries and salivary characteristics among type 1 diabetic Saudi children. J Dent Sci. 2022 Oct;17(4):1634-1639. doi: 10.1016/j.jds.2022.03.010. Epub 2022 Apr 6. PMID 36299323